CLINICAL TRIAL: NCT06587100
Title: Wearable Activity Tracking to Curb Hospitalizations (WATCH)
Brief Title: Wearable Activity Tracking to Curb Hospitalizations
Acronym: WATCH
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23722; NCI-2024-06762 (Registry Identifier: NCI Clinical Trial Reporting Program (CTRP)); R01CA277782 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Neoplasm; Malignant Solid Neoplasm; Lymphatic System Neoplasm
Keywords: Activity tracking; Hospitalization prevention; Artificial Intelligence (AI) modelling
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Group I: Fitbit only: Participants receive Fitbit device while undergoing non-interventional, standard of care, radiation therapy.
  Interventions: Device: Fitbit
- Observational Group II: Fitbit + Apple HealthKit: Participants receive Fitbit device and will utilize personal Apple HealthKit-based devices (iPhone, Apple Watch, etc.) to concurrently contribute Apple HealthKit-based data while undergoing non-interventional, standard of care, radiation therapy.
  Interventions: Device: Fitbit; Device: Apple HealthKit-based devices

INTERVENTIONS:
Device: Fitbit — Participants will wear Fitbit device
  Other Names: Wearable Activity Tracker
Device: Apple HealthKit-based devices — Participants will wear personal device and share data with study team.
  Other Names: iPhone; Apple watch
  Groups: Observational Group II: Fitbit + Apple HealthKit

SUMMARY:
This study is being done to collect patient generated health data to predict the risk of patients needing emergency department visits or hospitalization before, during. and after receiving radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Validate a previously developed step-count model for predicting all-cause acute care (pooled across all devices).

SECONDARY OBJECTIVES:

I. Validate a previously developed model for predicting each ED visits or hospitalizations during external beam RT using continuous step counts before, during, and after treatment.

II. Validate the previously developed step-count model for predicting all-cause acute care for each of the two different device platforms.

III. Validate concordance of step counts across each of the device's platforms in the Apple group.

IV. Validate the previously developed SHIELD-RT Electronic health record (EHR)-based model for predicting unplanned acute care (ED visit or hospitalization).

EXPLORATORY OBJECTIVES:

I. Refinement of the pre-existing models(step count and SHIELD-RT). II. Evaluate association between wearables collected parameters, EHR-based variables, and acute care events.

III. Develop and validate a multi-modal predictive model for predicting acute care.

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 groups.

* GROUP I: Participants receive Fitbit device and undergo non-interventional, standard of care, radiation therapy.
* GROUP II: Participants receive Fitbit device and utilize their own personal Apple HealthKit-based device and undergo non-interventional, standard of care, radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Able to understand study procedures and to comply with them for the entire length of the study.
* Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
* Diagnosis of invasive malignancy.
* Able to ambulate independently (without the assistance of a cane or walker).
* Planned treatment with fractionated external beam radiotherapy over at least 5 days (no fractional requirement).
* Not a previous participant on this protocol for subsequent courses.

Exclusion Criteria:

* Participants bound to a wheelchair.
* Participants unable to ambulate independently (needing assistance of cane or walker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing non-interventional, standard of care, radiotherapy (RT) at UCSF Department of Radiation Oncology
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUC-ROC) of the step count model | Up to 3 years
  The AUC-ROC of the step count model will measure the performance of a classification model by plotting the rate of true positives against false positives, and the score ranges from 0 - 1. The higher the AUC, the better the model's performance at distinguishing between the positive and negative classes. The AUC-ROC will be reported including both estimates and confidence intervals. All models will be reported per up-to-date guidelines, such as Minimum Information about Clinical Artificial Intelligence Modeling (MI-CLAIM) and Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD). The performance metrics will only be calculated with respect to first acute care event.
Calculation of a Brier Score | Up to 3 years
  The Brier Score is a strictly proper score function or strictly proper scoring rule that measures the accuracy of probabilistic predictions. A Brier Score can take on any value between 0 and 1, with 0 being the best score achievable and 1 being the worst score achievable. The lower the Brier Score, the more accurate the prediction(s). The score will be reported including both estimates and confidence intervals. All models will be reported per up-to-date guidelines, such as MI-CLAIM and TRIPOD. The performance metrics will only be calculated with respect to first acute care event.
Calculation of Log-Loss Score | Up to 3 years
  Logarithmic loss indicates how close a prediction probability comes to the actual/corresponding true value. The Log-Loss Score can take on any value between 0 and 1. The more the predicted probability diverges from the actual value, the higher is the log-loss value. The log-loss value will be reported including both estimates and confidence intervals. All models will be reported per up-to-date guidelines, such as MI-CLAIM and TRIPOD. The performance metrics will only be calculated with respect to first acute care event.
Area Under the Precision-Recall Curves (AUCPR) | Up to 3 years
  The area under the precision-recall curve (AUCPR) is a single number summary of the information in the precision-recall (PR) curve. It represents the tradeoff between precision and recall for different thresholds, where high AUCPR indicates both high recall and high precision. The AUCPR will be reported including both estimates and confidence intervals. All models will be reported per up-to-date guidelines, such as MI-CLAIM and TRIPOD. The performance metrics will only be calculated with respect to first acute care event.

SECONDARY OUTCOMES:
AUC-ROC for composite acute care | Up to 3 years
  The AUC-ROC will be used to validate a previously developed model in the primary endpoint for predicting each ED visits or hospitalizations during external beam RT using continuous step counts before, during, and after treatment.
Area under the receiver operating characteristic curve (AUC-ROC) for all cause acute care by group | Up to 3 years
  The AUC-ROC will be used to validate the previously developed step-count model in the primary endpoint for predicting all-cause acute care for each of the two different device platforms.
Mean squared error (MSE) | Up to 3 years
  The MSE will be used to validate concordance of step counts across each of the device's platforms in the Apple group. Mean Squared Error (MSE) is a fundamental concept in statistics and machine learning in assessing the accuracy of the predictive models which measures the average squared difference between predicted values and the actual values in the dataset.
Area under the receiver operating characteristic curve (AUC-ROC) for the composite acute care endpoint.. | Up to 3 years
  Validate the previously developed SHIELD-RT EHR-based model for predicting unplanned acute care (ED visit or hospitalization) to discover additional variables which may be predictors not previously included.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Hong, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No